CLINICAL TRIAL: NCT06592768
Title: A Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of Briquilimab in Participants With Allergic Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision - terminated due to changes in company priorities and not related to safety concerns.
Sponsor: Jasper Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JSP-CP-012; 2024-516164-28-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Allergic Asthma
Keywords: Asthma; Allergy; Chronic Disease; Lung Function; Exacerbation; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases
MeSH Terms: conditions — Asthma; Hypersensitivity; Chronic Disease; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: This study is designed as a double-blind, placebo-controlled, parallel-group, randomized, study to evaluate the safety and efficacy of briquilimab on allergen-induced asthmatic airway responses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator
- Briquilimab (Experimental)
  Interventions: Drug: Briquilimab

INTERVENTIONS:
Drug: Briquilimab — Subcutaneous Administration
  Other Names: JSP191
  Arms: Briquilimab
Other: Placebo Comparator — Subcutaneous Administration
  Arms: Placebo

SUMMARY:
Study JSP-CP-012 is designed as a proof of concept, parallel-group, single dose, double blind, placebo-controlled study using an allergen challenge model. A single dose proof of concept approach at a dose level shown to be biologically active should inform the impact of briquilimab on allergic asthma as compared to placebo while minimizing exposure to participants, in a new indication.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age; stable, allergic asthma; history of episodic wheeze and shortness of breath; forced expiratory volume in 1 second (FEV1) at baseline at least 70% of the predicted value; able to comprehend and follow all required study procedures; willing and able to sign an informed consent form; positive methacholine challenge at baseline (concentration of methacholine causing 20% decrease in FEV1 [PC20] PC20 ≤ 16 mg/mL or PD20 equivalent to ≤400µg); and positive skin-prick test and positive allergen-induced early and late airway bronchoconstriction to common aeroallergens.

Exclusion Criteria:

* Worsening of asthma or respiratory infection in the preceding 6 weeks; lung disease other than allergic asthma; prior treatment with a c-Kit inhibiting therapy; anaphylaxis to any parenterally administered biologics; use of asthma medications (note: intermittent doses of short-acting β2-agonist are allowed once weekly for relief of symptoms but prophylactic use for exercise is allowed as-needed); pregnant or lactating women; and women actively seeking pregnancy or who are not using adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of briquilimab in mild-to-moderate asthmatic participants | From signing the informed consent form (ICF) through end of trial (EOT) visit (up to 4.5 months)
  Incidence and/or severity of AEs, treatmentemergent adverse events (TEAEs), SAEs, AEIs, and AEs leading to discontinuation.
  Incidence of clinically significant abnormal laboratory values and vital signs.
To compare the effect of treatment with briquilimab vs placebo on the allergen-induced LAR | 3-7 hours after allergen challenge between Briquilimab and Placebo at week 6
  Allergen-induced LAR will be measured by maximum percentage fall in FEV1 during the period 3-7 hours after the allergen challenge and compared between briquilimab and placebo at week 6.
To compare the effect of treatment with briquilimab vs placebo on the allergen-induced LAR | 3-7 hours after allergen challenge between Briquilimab and Placebo at week 6
  Allergen-induced LAR will be measured by area under the FEV1 time-response curve [AUC] during the period 3-7 hours after the allergen challenge and compared between briquilimab and placebo at week 6.

SECONDARY OUTCOMES:
To compare of the allergen-induced early asthmatic response (EAR) between briquilimab and placebo. | 0-2 hours after the allergen challenge and compared briquilimab and placebo at week 6
  Allergen-induced EAR will be measured by maximum percentage fall in FEV1 during the period 0-2 hours after the allergen challenge and compared briquilimab and placebo at week 6.
To compare of the allergen-induced early asthmatic response (EAR) between briquilimab and placebo. | 0-2 hours after the allergen challenge and compared briquilimab and placebo at week 6
  Allergen-induced EAR will be measured by area under the FEV1 time-response curve [AUC] during the period 0-2 hours after the allergen challenge and compared briquilimab and placebo at week 6.
Comparison of allergen-induced inflammatory mediators at 7h and 24h post allergen, between briquilimab and placebo | 7 hours and 24 hours after the allergen challenge, compared between briquilimab and placebo at week 6.
  Changes from pre-allergen challenge sputum inflammatory mediators to 7 hours and 24 hours after the allergen challenge, compared between briquilimab and placebo at week 6.
Comparison of the allergen-induced shift in AHR to methacholine at 24 hours after the allergen challenge, between briquilimab and placebo. | 24 hours after the allergen challenge compared between briquilimab and placebo at week 6.
  Changes from pre-allergen challenge AHR to 24 hours after the allergen challenge assessed by methacholine PD20, and compared between briquilimab and placebo at week 6.
Comparison of the allergen-induced changes in sputum leukocytes at 7h and 24h post allergen challenge, between the briquilimab and placebo. | 7 hours and 24 hours after the allergen challenge, compared between briquilimab at week 6. and placebo.
  Changes from pre-allergen challenge sputum leukocytes to 7 hours and 24 hours after the allergen challenge, compared between briquilimab and placebo at week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Jasper Therapeutics
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - University of Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No